CLINICAL TRIAL: NCT03525496
Title: Interest of Challenge Tests for Diagnosis of Immediate Hypersensitivity Against Iodinated Contrast Agents
Acronym: DHIODE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01Obs-CHRMT
Record Dates: First submitted 2018-04-24; First posted 2018-05-15 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-04

CONDITIONS: Allergic Reaction
Keywords: Iodinated contrast agents; Immediate hypersensitivity reactions; Reintroduction tests
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Iodinated contrast agents (ICA) are widely used in medical imaging. They provide however a risk of immediate hypersensitivity reactions (IHS). The risk of anaphylactic shock is estimated at 1/100 000 injections. Nevertheless, for safety reasons and to limit undesirable effects, the reintroduction tests are not conducted along similar lines to throughout scan or arteriography. Moreover, reintroduction protocols are actually not standardized, in terms of injected volume and doses progression. It should be evaluated the relevance of the reintroduction tests with injection of a low volume and ensure the absence of reaction during the ICA injections Under real conditions.

The investigators are assuming that the realization of a provocation test by intravenous reintroduction with a reduced dose of ICA improves the predictive value of IHS in comparison with only cutaneous tests.

DETAILED DESCRIPTION:
The main objective of this study will be to estimate the negative predictive value of the combination of cutaneous tests and provocation test by intravenous reintroduction in the IHS to iodinated contrast agents.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Having suffered single-blind reintroduction
* Having benefited from cutaneous tests and ICA reintroduction test in the framework of IHS

Exclusion Criteria:

* Patient with delayed hypersensitivity
* Opposed to use data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patient who had an iodinated contrast agents reintroduction test
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of immediate hypersensitivity reactions | Day 1
  Occurrence of immediate hypersensitivity reactions after an injection of ICA

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz-Thionville, Metz, Moselle, France